CLINICAL TRIAL: NCT02973321
Title: A 26-Week Randomized, Double-blind, Placebo-controlled, Dose-ranging Phase 2 Study to Assess the Safety and Efficacy of SAR425899 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Safety and Efficacy of SAR425899 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI13940; 2016-001328-77 (EudraCT Number); U1111-1179-4786 (Other: UTN)
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — SAR425899; Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo (for SAR425899) subcutaneous (SC) injection once daily (QD) from Week 1 to Week 26, matching 3 SAR425899 dose levels of 0.12 mg, 0.16 mg and 0.20 mg.
  Interventions: Drug: Placebo; Drug: Metformin
- SAR425899 0.12 mg (Experimental): SAR425899 SC injection QD at maintenance dose of 0.12 mg for 25 weeks (Week 2 to Week 26) following 1 week dose increase step (0.06 mg at Week 1).
  Interventions: Drug: SAR425899; Drug: Metformin
- SAR425899 0.16 mg (Experimental): SAR425899 SC injection QD at maintenance dose of 0.16 mg for 24 weeks (Week 3 to Week 26) following 2 weeks dose increase step (0.06 mg at Week 1 and 0.12 mg at Week 2).
  Interventions: Drug: SAR425899; Drug: Metformin
- SAR425899 0.20 mg (Experimental): SAR425899 SC injection QD at maintenance dose of 0.20 mg for 23 weeks (Week 4 to Week 26) following 3 weeks dose increase step (0.06 mg at Week 1, 0.12 mg at Week 2 and 0.16 mg at Week 3).
  Interventions: Drug: SAR425899; Drug: Metformin
- Liraglutide (Active Comparator): Liraglutide SC injection QD at maintenance dose of 1.8 mg for 24 weeks (Week 3 to Week 26) following 2 weeks dose increase steps (0.6 mg daily at Week 1 and by 1.2 mg daily at Week 2).
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: SAR425899 — Self-administered by SC injection using a solution for injection in cartridge.
  Arms: SAR425899 0.12 mg; SAR425899 0.16 mg; SAR425899 0.20 mg
Drug: Placebo — Self-administered by SC injection using a solution for injection in cartridge.
  Arms: Placebo
Drug: Liraglutide — Self-administered by SC injection using a pre-filled pen.
  Other Names: Victoza
  Arms: Liraglutide
Drug: Metformin — Orally administered at a stable dose , >=1500 mg daily stable dose or maximal tolerated dose.

SUMMARY:
Primary Objective:

The primary objective of this study was to assess the dose-response relationship of SAR425899 versus placebo in terms of glycemic control as measured by the change in glycosylated hemoglobin (HbA1c).

Secondary Objectives:

* To assess the effect of SAR425899 on body weight.
* To assess the safety and immunogenicity profile of SAR425899, including assessment of the heart rate (HR) change by electrocardiogram (ECG) and Holter monitor.
* To assess the proportion of participants achieving predefined HbA1c targets of <7% and <6.5% as well as the proportion of participants achieving >=5% and >=10% body weight loss.
* To assess the effect of once daily dosing of SAR425899 on additional parameters of glycemic control and lipid metabolism.
* To assess the effect of once daily dosing of SAR425899 on additional pharmacodynamic (PD) biomarkers.
* To assess the pharmacokinetic (PK) profile and parameters of SAR425899, inter-individual and inter-occasion variability in PK parameters using a population PK approach.

DETAILED DESCRIPTION:
The total study duration will be approximately 30 weeks, consisting of 3 weeks screening period at the site, a 26 weeks treatment period, and 3 days post treatment follow up period.

ELIGIBILITY:
Inclusion criteria :

* Participants with type-2 diabetes mellitus (T2DM) for at least 3 months before the screening visit.
* On diet/exercise and/or treatment with metformin (stable dose of ≥1500 mg/day or maximal tolerated dose) for at least 3 months prior to screening.
* Signed informed consent.

Exclusion criteria:

* At screening, participant's age < legal age of adulthood and >80 years.
* Glycated hemoglobin at screening visit <7.0% or >10.0%.
* Body mass index (BMI) <25 kg/m^2 or >45.0 kg/m^2.
* Pregnant or lactating women.
* Women of childbearing potential (WOCBP) not protected by highly-effective method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy.
* Diagnosis of type 1 diabetes mellitus.
* Fasting plasma glucose of >15 mmol/L (270 mg/dL) measured by the central laboratory at screening (Visit 1), and confirmed (>15 mmol/L [270 mg/dL]) by a repeat test before randomization.
* Treatment with glucose-lowering agents(s) other than metformin, currently or within the 3 months prior to screening.
* Previous insulin use, except for episode(s) of short-term treatment (≤15 consecutive days) for intercurrent illness or pregnancy, or use of insulin within the last 6 months.
* Contraindication(s) to metformin use.
* Contraindication(s) to liraglutide use.
* Significant change in body weight in the 3 months before screening.
* Poorly controlled hypertension (a resting systolic blood pressure (SBP) >160 mm Hg and/or diastolic blood pressure (DBP) >95 mm Hg at screening).
* History of long QT syndrome and/or QTc more than 450 ms at screening visit.
* History of pancreatitis or pancreatectomy.
* History of weight loss surgery.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predispose to MTC.
* Any prior exposure to drugs belonging to the class of glucagon-like peptide-1 (GLP-1) receptor agonists/GLP-1 analogs.
* Contraindications or known hypersensitivity reaction to glucagon.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (59):
- United States (23):
  - Investigational Site Number 8400028, Sheffield, Alabama
  - Investigational Site Number 8400002, Huntington Park, California
  - Investigational Site Number 8400024, Los Angeles, California
  - Investigational Site Number 8400001, Los Angeles, California
  - Investigational Site Number 8400012, Port Hueneme, California
  - Investigational Site Number 8400027, Denver, Colorado
  - Investigational Site Number 8400025, Miami, Florida
  - Investigational Site Number 8400007, Palm Harbor, Florida
  - Investigational Site Number 8400013, Chicago, Illinois
  - Investigational Site Number 8400016, Wichita, Kansas
  - Investigational Site Number 8400023, Wichita, Kansas
  - Investigational Site Number 8400018, New Orleans, Louisiana
  - Investigational Site Number 8400019, Rockville, Maryland
  - Investigational Site Number 8400014, Flint, Michigan
  - Investigational Site Number 8400003, Troy, Michigan
  - Investigational Site Number 8400020, Linden, New Jersey
  - Investigational Site Number 8400022, New York, New York
  - Investigational Site Number 8400005, Fargo, North Dakota
  - Investigational Site Number 8400004, Austin, Texas
  - Investigational Site Number 8400006, Dallas, Texas
  - Investigational Site Number 8400021, Houston, Texas
  - Investigational Site Number 8400026, San Antonio, Texas
  - Investigational Site Number 8400017, Sugar Land, Texas
- Canada (5):
  - Investigational Site Number 1240008, Québec
  - Investigational Site Number 1240005, Sainte-Foy
  - Investigational Site Number 1240002, Sherbrooke
  - Investigational Site Number 1240001, Toronto
  - Investigational Site Number 1240003, Vancouver
- Czechia (4):
  - Investigational Site Number 2030003, České Budějovice
  - Investigational Site Number 2030001, Krnov
  - Investigational Site Number 2030004, Praha 10 - Uhrineves
  - Investigational Site Number 2030002, Praha 9 - Klanovice
- Germany (3):
  - Investigational Site Number 2760003, Berlin
  - Investigational Site Number 2760001, Dresden
  - Investigational Site Number 2760006, Hohenmölsen
- Hungary (6):
  - Investigational Site Number 3480001, Balatonfüred
  - Investigational Site Number 3480002, Budapest
  - Investigational Site Number 3480008, Budapest
  - Investigational Site Number 3480005, Budapest
  - Investigational Site Number 3480006, Budapest
  - Investigational Site Number 3480007, Budapest
- Mexico (5):
  - Investigational Site Number 4840004, Actopan
  - Investigational Site Number 4840001, Guadalajara
  - Investigational Site Number 4840003, Guadalajara
  - Investigational Site Number 4840002, Monterrey
  - Investigational Site Number 4840006, San Juan del Río
- Russia (5):
  - Investigational Site Number 6430002, Saint Petersburg
  - Investigational Site Number 6430004, Saint Petersburg
  - Investigational Site Number 6430001, Saint Petersburg
  - Investigational Site Number 6430003, Saratov
  - Investigational Site Number 6430005, Voronezh
- Spain (8):
  - Investigational Site Number 7240001, A Coruña
  - Investigational Site Number 7240005, Barcelona
  - Investigational Site Number 7240007, Ferrol
  - Investigational Site Number 7240006, Las Palmas de Gran Canaria
  - Investigational Site Number 7240002, Madrid
  - Investigational Site Number 7240003, Málaga
  - Investigational Site Number 7240004, Málaga
  - Investigational Site Number 7240008, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Schiavon M, Visentin R, Gobel B, Riz M, Cobelli C, Klabunde T, Dalla Man C. Improved postprandial glucose metabolism in type 2 diabetes by the dual glucagon-like peptide-1/glucagon receptor agonist SAR425899 in comparison with liraglutide. Diabetes Obes Metab. 2021 Aug;23(8):1795-1805. doi: 10.1111/dom.14394. Epub 2021 May 5. PMID 33822469
- [Derived] Gater A, Reaney M, Findley A, Brun-Strang C, Burrows K, Nguyen-Pascal ML, Roborel de Climens A. Development and First Use of the Patient's Qualitative Assessment of Treatment (PQAT) Questionnaire in Type 2 Diabetes Mellitus to Explore Individualised Benefit-Harm of Drugs Received During Clinical Studies. Drug Saf. 2020 Feb;43(2):119-134. doi: 10.1007/s40264-019-00877-4. PMID 31679129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 59 centers in 8 countries. A total of 539 participants were screened between 2 December 2016 and 2 June 2017, of whom, 245 participants were screen failures. Screen failures were mainly due to exclusion criteria met. The study was double-blind for SAR425899 vs placebo and open-label for active comparator liraglutide.
Pre-assignment Details: Total of 294 participants were randomized using interactive response technology, however 2 participants were screened failures and were randomized by error in liraglutide and SAR425899 0.20 mg groups, therefore a total of 296 participants were randomized and treated in study. Randomization was stratified by glycosylated hemoglobin(HbA1c) at screening visit(<8% vs >=8%) and body mass index (BMI)(<35.0 kg/m^2 vs >=35.0kg/m^2) at Day 1(start of investigational medicinal product[IMP]administration).
Period: Overall Study
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Started | 33 | 66 | 66 | 64 | 67
Completed | 32 | 51 | 52 | 48 | 62
Not Completed | 1 | 15 | 14 | 16 | 5
Not completed — Other than specified | 0 | 5 | 3 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 10 | 11 | 13 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Placebo: Placebo (for SAR425899) SC injection QD from Week 1 to Week 26, matching 3 SAR425899 dose levels of 0.12 mg, 0.16 mg and 0.20 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide | Total
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (9.3) | 56.8 (9.0) | 54.5 (10.1) | 55.0 (10.4) | 56.1 (11.4) | 55.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 29 | 35 | 28 | 36 | 143
  Male | 18 | 37 | 31 | 36 | 31 | 153
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian/Oriental | 0 | 1 | 1 | 2 | 1 | 5
  Black | 2 | 6 | 6 | 2 | 4 | 20
  White | 31 | 59 | 59 | 59 | 61 | 269
  Other | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 15 | 19 | 25 | 28 | 13 | 100
  Non Hispanic | 18 | 47 | 41 | 36 | 54 | 196
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.07 (4.41) | 33.67 (5.37) | 34.23 (4.68) | 33.63 (4.35) | 34.23 (5.51) | 33.74 (4.96)
Baseline HbA1c [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.04 (0.86) | 7.97 (0.88) | 7.99 (0.85) | 8.14 (0.94) | 8.11 (0.86) | 8.05 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Week 26
Description: Change in HbA1c was calculated by subtracting baseline value from Week 26 value. Missing post-baseline values were imputed by placebo control-based multiple imputation (MI) method under the missing not at random framework.
Time Frame: Baseline, Week 26
Population: Analysis was performed on Intent-to-treat (ITT) population which included all randomized participants, irrespective of compliance with the study protocol and procedures.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
percentage of HbA1c | -0.663 (0.169) | -1.517 (0.137) | -1.618 (0.133) | -1.562 (0.131) | -1.312 (0.118)
Statistical Analysis 1: Comparison: Placebo vs SAR425899 0.12 mg vs SAR425899 0.16 mg vs SAR425899 0.20 mg; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Visit 4 (Day 1) BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline HbA1c as a covariate. Overall 1st trend test based on a contrast with coefficients of +3, +1, -1, -3 and 0 for SAR425899 0.20 mg, 0.16 mg, 0.12 mg, placebo and liraglutide. Here it is test 1 of testing order; Test type: Other — The overall Type 1 error for multiple comparisons of the HbA1c and body weight was controlled by a Hierarchical testing procedure. Testing was performed in following sequence: 1. 1st trend test for HbA1c, 2. 1st trend test for body weight, 3. 2nd trend test for HbA1c, 4. 2nd trend test for body weight, 5. 3rd trend test for HbA1c, 6. 3rd trend test for body weight; p < 0.0001, ANCOVA — Hierarchical testing procedure continued only, if the previous comparison was statistically significant. Threshold for significance at 0.05 level; 1st trend test
Statistical Analysis 2: Comparison: Placebo vs SAR425899 0.16 mg; Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Visit 4 (Day 1) BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline HbA1c as a covariate. Second Trend test based on a contrast with coefficients of 0, +1, 0, -1 and 0 for SAR425899 0.20 mg, 0.16 mg, 0.12 mg, placebo and liraglutide, respectively. Here, it is test no. 3 of hierarchical testing sequence; Test type: Other — Hierarchical testing procedure continued only, if the previous comparison was statistically significant; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; 2nd Trend test; LS Mean difference = -0.956, 95% CI 2-sided [-1.359 to -0.552], Standard Error of Mean 0.206
Statistical Analysis 3: Comparison: Placebo vs SAR425899 0.12 mg; Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Visit 4 (Day 1) BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline HbA1c as a covariate. Third Trend test based on a contrast with coefficients of 0, 0, +1, -1 and 0 for SAR425899 0.20 mg, 0.16 mg, 0.12 mg, placebo and liraglutide, respectively. Here, it is test no. 5 of hierarchical testing sequence; Test type: Other — Hierarchical testing procedure continued only, if the previous comparison was statistically significant; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; 3rd Trend test; LS Mean difference = -0.854, 95% CI 2-sided [-1.264 to -0.444], Standard Error of Mean 0.209

2. Secondary Outcome: Mean Change From Baseline in Body Weight to Week 26
Description: Change in body weight was calculated by subtracting baseline value from Week 26 value. Missing post- baseline values were imputed by placebo control-based MI method under the missing not at random framework.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
Kg | -1.759 (0.734) | -4.276 (0.564) | -5.330 (0.549) | -4.407 (0.559) | -4.590 (0.521)
Statistical Analysis 1: Comparison: Placebo vs SAR425899 0.12 mg vs SAR425899 0.16 mg vs SAR425899 0.20 mg; Placebo, SAR425899 0.12,0.16,0.20 mg: Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Day 1 BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline body weight as a covariate. Here, it is test no. 2 of hierarchical testing sequence; Test type: Other — Hierarchical testing procedure continued only, if the previous comparison was statistically significant; p = 0.0012, ANCOVA — Threshold for significance at 0.05 level; 1st Trend test
Statistical Analysis 2: Comparison: Placebo vs SAR425899 0.16 mg; SAR425899 0.16 mg vs Placebo: Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Day 1 BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline body weight as a covariate. Here, it is test no. 4 of hierarchical testing sequence; Test type: Other — Hierarchical testing procedure continued only, if the previous comparison was statistically significant; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; 2nd Trend test; LS Mean difference = -3.57, 95% CI 2-sided [-5.309 to -1.832], Standard Error of Mean 0.887
Statistical Analysis 3: Comparison: Placebo vs SAR425899 0.12 mg; 3rd Trend Test: SAR425899 0.12 mg vs Placebo: Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c value (<8, >=8 %), randomization strata of Day 1 BMI (<35.0 kg/m^2, >=35.0 kg/m^2), and country as fixed effects and baseline body weight as a covariate. Here, it is test no. 6 of hierarchical testing sequence; Test type: Other — Hierarchical testing procedure continued only, if the previous comparison was statistically significant; p = 0.0047, ANCOVA — Threshold for significance at 0.05 level; 3rd Trend test; LS Mean difference = -2.517, 95% CI 2-sided [-4.264 to -0.77], Standard Error of Mean 0.891

3. Secondary Outcome: Percentage of Participants Reached HbA1c Target of <6.5% or <7% at Week 26
Description: The analysis included assessment collected during the study, including those obtained after IMP discontinuation or introduction of rescue therapy. Participants with no measurement at Week 26 were treated as non-responders.
Time Frame: Week 26
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
percentage of participants
  Participants with HbA1c Target of <6.5% | 12.1 | 47.0 | 51.5 | 48.4 | 44.8
  Participants with HbA1c Target of <7% | 36.4 | 66.7 | 68.2 | 65.6 | 67.2

4. Secondary Outcome: Percentage of Participants Achieving >=5% or >=10% Body Weight Loss at Week 26
Description: as for outcome 3
Time Frame: Week 26
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
percentage of participants
  Participants Achieving >=5% Body Weight Loss | 3.0 | 33.3 | 45.5 | 35.9 | 40.3
  Participants Achieving >=10% Body Weight Loss | 0.0 | 12.1 | 13.6 | 15.6 | 9.0

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Week 26
Description: Change in FPG was calculated by subtracting baseline value from Week 26 value. Missing post-baseline values were imputed by placebo control-based MI method under the missing not at random framework.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
mmol/L | -0.931 (0.394) | -2.408 (0.308) | -2.548 (0.301) | -2.318 (0.312) | -2.124 (0.280)

6. Secondary Outcome: Change From Baseline in Average 7 Point Self-Monitoring Plasma Glucose (SMPG) to Week 26
Description: Change in 7-point SMPG profile from baseline to Week 26 was assessed by summary statistics. 7-point SMPG profiles were measured at the following 7 points at each visit (Baseline, and Week 26): pre-prandial and 2 hours postprandial for breakfast, lunch, dinner and at bedtime. Two hours postprandial (breakfast, lunch and dinner) is defined as 2 hours after the start of the meal.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Overall number of participants analyzed = participants with at least 1 baseline and 1 post-baseline SMPG assessment during 26 week treatment period.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 21 | 40 | 43 | 44 | 49
mmol/L | -1.82 (3.11) | -2.86 (2.62) | -2.63 (2.70) | -2.49 (3.18) | -2.21 (2.23)

7. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy
Description: Rescue medication was introduced in case FPG or HbA1c values were above pre-defined thresholds, and if no reasons were found for insufficient glucose control, and appropriate action failed to decrease FPG / HbA1c under the threshold values (from baseline to Week 8: FPG >270 mg/dL 15.0 mmol/L, from Week 8 to Week 14: FPG >13.3 mmol/L, and from Week 14 to Week 26: FPG >11.1 mmol/L or HbA1c>8%). The choice of rescue therapy was at the Investigator's discretion with the exception of using glucagon-like peptide-1 receptor (GLP-1R) agonists or dipeptidyl peptidase 4 (DPP4) inhibitors.
Time Frame: Baseline up to 26 weeks
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
percentage of participants | 18.2 | 0.0 | 1.5 | 3.1 | 6.0

8. Secondary Outcome: Change From Baseline in Beta-Cell Function to Week 26
Description: Beta-cell function was assessed by homeostatic model assessment (HOMA)-beta, derived from FPG and fasting plasma insulin (FPI). HOMA-beta was derived from FPG and FPI as (20*FPI [micro units/milliliter]) divided by (FPG [mmol/L] minus 3.5). Change was calculated for HOMA-beta by subtracting the Baseline value from Week 26 value*100.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of normal beta cells function
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
percentage of normal beta cells function | 15.025 (19.785) | 26.768 (15.833) | 31.122 (16.467) | 17.932 (14.397) | 27.263 (13.234)

9. Secondary Outcome: Change From Baseline in Insulin Resistance to Week 26
Description: Insulin Resistance was assessed by homeostasis model assessment for insulin resistance (HOMA-IR), derived from FPG and FPI. HOMA-IR was derived from FPG and FPI as (FPI [micro units per milliliter] * FPG [mmol/L]) divided by 22.5. Change was calculated for HOMA-beta by subtracting the Baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: HOMA-IR Index
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
HOMA-IR Index | -1.315 (0.865) | -1.244 (0.670) | -2.233 (0.664) | -2.324 (0.649) | -1.405 (0.613)

10. Secondary Outcome: Change From Baseline in Pharmacodynamic Biomarkers to Week 26 - Waist and Hip Circumferences
Description: Waist circumference was measured at the midpoint between the lower margin of the least palpable rib and the top of the iliac crest, using a stretch-resistant tape providing a constant 100 gm tension. Hip circumference was measured around the widest portion of the buttocks, with the tape parallel to the floor. Each measurement was repeated twice; if the measurements were within 1 cm of one another, the average was calculated, and if the difference exceeded 1 cm, the measurements were repeated.
Time Frame: Baseline,Week 26
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Placebo | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
Number analyzed (Participants) | 33 | 66 | 66 | 64 | 67
cm
  Waist Circumference | -2.0 (0.75) | -5.3 (1.34) | -2.3 (1.61) | -3.2 (0.66) | -4.0 (2.03)
  Hip Circumference | -1.42 (0.781) | -4.46 (1.378) | -1.97 (1.572) | -4.09 (0.945) | -2.56 (1.513)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form until 3 days after last treatment administration (Day 185).
Description: Reported AEs were treatment-emergent AEs that is AEs that developed/worsened or became serious during the 26-week'treatment period' (Treatment period was defined as time from the first injection of IMP up to last injection of IMP + 3 days). AE data was planned to be reported based on the dose received starting at Week 8 when adjustment of dose was not allowed (or randomized treatment arm if participant discontinued before Week 8).
Groups:
- SAR425899 0.06 mg: Participants who were originally randomized to SAR425899 treatment groups and received 0.06 mg QD at Week 8.
- SAR425899 0.12 mg: Participants who were originally randomized to SAR425899 treatment groups and received 0.12 mg QD at Week 8, or participants randomized to SAR425899 0.12 mg treatment group and discontinued the study before Week 8.
- SAR425899 0.16 mg: Participants who were originally randomized to SAR425899 treatment groups and received 0.16 mg QD at Week 8, or participants randomized to SAR425899 0.16 mg treatment group and discontinued the study before Week 8.
- SAR425899 0.20 mg: Participants who were originally randomized to SAR425899 treatment groups and received 0.20 mg QD at Week 8, or participants randomized to SAR425899 0.20 mg treatment group and discontinued the study before Week 8.
- Liraglutide: Participants randomized to and received Liraglutide treatment were included in the Liraglutide treatment arm regardless of dose amount participants received.
Arm/Group | Placebo | SAR425899 0.06 mg | SAR425899 0.12 mg | SAR425899 0.16 mg | SAR425899 0.20 mg | Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/18 | 0/72 | 0/59 | 0/47 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/33 | 2/18 | 3/72 | 1/59 | 2/47 | 2/67
Other Adverse Events (participants affected / at risk) | 10/33 | 18/18 | 49/72 | 45/59 | 34/47 | 34/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | SAR425899 0.06 mg (N=18) | SAR425899 0.12 mg (N=72) | SAR425899 0.16 mg (N=59) | SAR425899 0.20 mg (N=47) | Liraglutide (N=67)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases To Adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | SAR425899 0.06 mg (N=18) | SAR425899 0.12 mg (N=72) | SAR425899 0.16 mg (N=59) | SAR425899 0.20 mg (N=47) | Liraglutide (N=67)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 1 (1) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 5 (6) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (5) | 2 (2) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5) | 6 (6) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 7 (10) | 15 (23) | 11 (16) | 9 (14) | 8 (10)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 6 (8) | 13 (14) | 4 (4) | 3 (4) | 5 (5)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Gingival Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 13 (22) | 33 (45) | 33 (41) | 26 (36) | 21 (25)
Pyloric Sphincter Insufficiency (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 10 (17) | 21 (32) | 14 (23) | 17 (24) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 3 (3)
Injection Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (4) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 4 (4) | 5 (5) | 4 (4) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 5 (5) | 1 (1) | 1 (2) | 3 (3)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT02973321/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT02973321/SAP_001.pdf